CLINICAL TRIAL: NCT01092936
Title: Italian Validation of the Revised MDS-Unified Parkinson's Disease Rating Scale
Acronym: IRIS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fondazione Neureca (Other)
Responsible Party: Dr. Linda Toscano, Fondazione NEURECA
Other Study IDs: IRIS
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson's Disease
Keywords: Comparative fit index; Movement Disorders' Society; Unified Parkinson's Disease Rating Scale
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Rating Scale administration — Movement Disorder Society_Unified Parkinson's Disease Rating Scale will be submitted to the patient (with the help of the caregiver) in a single visit lasting about 40 minutes.

SUMMARY:
The present study is part of an international program and deals with the translation and validation program for the Italian version of the MDS-UPDRS.

The program will be articulated in three steps:

* Phase I: translation and back-translation of the MDS-UPDRS in Italian (completed)
* Phase II: Cognitive testing. This step is aimed at a preliminary testing of a subset of potentially culturally sensitive items in a limited set of PD patients (approximately 10). Should this phase identify issues in the understanding and ease of use of some items a revised translation of some individual items might be envisaged.
* Phase III: large validation testing: this phase will involve 350 PD patients from 12-14 Italian PD centres.

The IRIS protocol deals with phase II and III of the program.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent;
* native Italian-speaking patients or either sex;
* patients suffering from Parkinson's disease ranging from mild to severe, based on clinical judgement;
* presence of a native Italian-speaking caregiver.

Exclusion Criteria:

* Patients with evidence of other central nervous system disorders;
* patients with a degree of depression or dementia which may prevent and/or affect ratings.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Native Italian-speaking PD patients ranging from mild to severe
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Phase II: To test the appropriateness of the Italian translation and clear understanding of potentially cultural-sensitive items. To refine the translation, if necessary, prior to validation testing. | 6 months
Phase III: the primary outcome of phase III is to confirm factorial analysis of the Italian version against the factor structure of the English version, by each of the four sections of the scale. | 6 months

SECONDARY OUTCOMES:
The secondary outcome is to determine the Differential Item Function (DIF) which will be run on items by gender, race , disease severity, education and age. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Barone, Prof., Principal Investigator — Universita' Federico II di Napoli; Maurizio Zibetti, Dr, Principal Investigator — Azienda Sanitaria Ospedaliera "San Giovanni Battista di Torino" Le Molinette; Angelo Antonini, Prof, Principal Investigator — Ospedale San Camillo IRCCS Venezia; Gianni Pezzoli, Prof, Principal Investigator — Istituti Clinici di Perfezionamento Milano; Michele Tinazzi, Prof, Principal Investigator — Azienda Ospedaliera Universitaria Integrata Verona - Policlinico G.Rossi; Giovanni Abbruzzese, Prof, Principal Investigator — Universita' di Genova; Ubaldo Bonuccelli, Prof, Principal Investigator — Universita' di Pisa; Giovanni Fabbrini, Dr, Principal Investigator — Universita' La Sapienza di Roma; Letterio Morgante, Prof, Principal Investigator — Azienda Ospedaliera Universitaria Policlinico G.Martino di Messina; Mario Zappia, Prof, Principal Investigator — Azienda Ospedaliero-Universitaria Policlinico Vittorio Emanuele di Catania; Alberto Albanese, Prof, Principal Investigator — Istituto Neurologico Carlo Besta di Milano; Claudio Pacchetti, Principal Investigator — Istituto Neurologico Nazionale Fondazione IRCCS "C. Mondino" di Pavia; Aldo Quattrone, Prof, Principal Investigator — Policlinico Universitario Mater Domini di Catanzaro; Giovanni Cossu, Dr, Principal Investigator — Azienda Ospedaliera "G. Brotzu" di Cagliari; Aroldo Rossi, Prof, Principal Investigator — Universita' degli Studi di Perugia; Paolo Martinelli, Prof, Principal Investigator — Universita' di Bologna
Locations (1):
- Universita' Federico II di Napoli, Napoli, Italy

REFERENCES:
- [Background] S. Fahn et al: The Unified Rating Scale for Parkinsonism. In Fahn, Marsden, Jenner, Teychenne eds.: Recent Developments in Parkinson's disease. N.J. Macmillan Healthcare Information: 153-63, 1987
- [Background] Movement Disorder Society Task Force on Rating Scales for Parkinson's Disease. The Unified Parkinson's Disease Rating Scale (UPDRS): status and recommendations. Mov Disord. 2003 Jul;18(7):738-50. doi: 10.1002/mds.10473. PMID 12815652
- [Background] Goetz CG, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stebbins GT, Stern MB, Tilley BC, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, Van Hilten JJ, LaPelle N. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Process, format, and clinimetric testing plan. Mov Disord. 2007 Jan;22(1):41-7. doi: 10.1002/mds.21198. PMID 17115387
- [Background] Goetz CG, Tilley BC, Shaftman SR, Stebbins GT, Fahn S, Martinez-Martin P, Poewe W, Sampaio C, Stern MB, Dodel R, Dubois B, Holloway R, Jankovic J, Kulisevsky J, Lang AE, Lees A, Leurgans S, LeWitt PA, Nyenhuis D, Olanow CW, Rascol O, Schrag A, Teresi JA, van Hilten JJ, LaPelle N; Movement Disorder Society UPDRS Revision Task Force. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord. 2008 Nov 15;23(15):2129-70. doi: 10.1002/mds.22340. PMID 19025984
- [Background] Pagonabarraga J, Kulisevsky J, Llebaria G, Garcia-Sanchez C, Pascual-Sedano B, Gironell A. Parkinson's disease-cognitive rating scale: a new cognitive scale specific for Parkinson's disease. Mov Disord. 2008 May 15;23(7):998-1005. doi: 10.1002/mds.22007. PMID 18381647
- See also: Related Info — http://www.movementdisorders.org